CLINICAL TRIAL: NCT03327857
Title: A Phase I Study of Neihulizumab (ALTB-168) in Patients With Steroid-refractory Acute Graft-versus-host Disease (SR-aGVHD) or Treatment-refractory Acute Graft-versus-host Disease (TR-aGVHD)
Brief Title: Neihulizumab (ALTB-168) in Patients With Steroid-refractory Acute Graft-versus-host Disease or Treatment-refractory Acute Graft-versus-host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AltruBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017.002.01
Record Dates: First submitted 2017-10-13; First posted 2017-11-01 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Steroid-refractory Acute Graft-versus-Host Disease; Treatment-refractory Acute Graft-versus-Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neihulizumab (ALTB-168) (Experimental): Intravenous doses of Neihulizumab (ALTB-168)
  Interventions: Biological: Neihulizumab (ALTB-168)

INTERVENTIONS:
Biological: Neihulizumab (ALTB-168) — Single dose phase: Patients will receive single dose of Neihulizumab based on the protocol escalation criteria.
  Multiple dose phase: Parients will receive weekly doses of Neihulizumab for 4 weeks.

SUMMARY:
A Phase I study to establish the pharmacokinetics, pharmacodynamics, safety and efficacy profiles of Neihulizumab in patients with steroid-refractory or treatment refractory acute graft-versus-host disease (SR/TR-aGVHD)

DETAILED DESCRIPTION:
Neihulizumab (ALTB-168) is an immune checkpoint agonist antibody that regulates T cell homeostasis. The unique mechanism of action provides a natural regulation of T cell homeostasis that induces cell death preferentially in late-stage activated T cells without affecting resting T cells and early-activated T cells. Because pathogenic T cells underlying the inflammatory conditions are usually in late-stage activated state, eliminating this population of cells can potentially result in controlling autoimmune inflammation of T cell associated diseases, such as GvHD.

ELIGIBILITY:
Inclusion Criteria (must meet all of the following criteria):

1. Patients must have clinical aGVHD and pathologic findings consistent with the diagnosis by biopsy of at least 1 involved site, and

   1. progressed after 3 days of treatment with methylprednisolone (MP) 2 mg/kg/day equivalent, or
   2. did not improve after 7 days of treatment with MP 2 mg/kg/day equivalent, or
   3. progressed to involve a new organ after treatment with MP 1 mg/kg/day equivalent for skin and upper gastrointestinal (GI) GVHD, or
   4. recurred during or after a steroid taper
2. For single dose phase: Patients must have erythematous manifestations of cutaneous aGVHD. Characteristics of the rash must indicate active inflammation (red coloration) as distinct from resolving inflammation (brown coloration).
3. For single dose phase: Providers and patients must be willing to defer new systemic or cutaneous topical treatment of aGVHD for at least 36 hr after administration of Neihulizumab.
4. Patient must give informed consent and sign an approved consent form prior to any study procedures.
5. Females of childbearing potential must have a negative pregnancy test result before enrollment. Males and females of childbearing potential must agree to use a highly effective method of birth control during the study for at least 30 days after enrollment in the study.

Exclusion Criteria (may not meet any of the following criteria):

1. For single dose phase: Prior administration of anti-lymphocyte globulin or anti- thymocyte globulin for treatment of aGVHD.
2. For multiple dose phase: Has received any systemic treatment in addition to corticosteroids for aGVHD.
3. Stage 4 lower GI GVHD, defined by the presence of ileus, severe abdominal pain, or overt GI bleeding.
4. Uncontrolled infections not responding to antimicrobial therapy or requiring intensive critical care or vasopressors.
5. Evidence of end-organ cytomegalovirus (CMV) or adenovirus infection.
6. Known to have adenovirus, or Epstein Barr virus (EBV) viremia from screening according to institutional standard practice. Patients receiving appropriate antiviral treatment for CMV, HHV6 or hepatitis viremia are eligible on a case-by-case basis.
7. HIV infection or a known HIV-related malignancy.
8. Tuberculosis, history of tuberculosis or a known positive Quantiferon test for tuberculosis.
9. Unplanned donor lymphocyte infusion (DLI) for residual or relapsed malignancy or mixed chimerism. DLI as part of the planned HCT protocol is allowed.
10. Known relapsed or progressive malignancy after transplant, posttransplant lymphoproliferative disease or any secondary malignancy diagnosed after HCT.
11. Absolute neutrophil count (ANC) <1000/mm3.
12. Total serum bilirubin concentration >3.0 mg/dL UNLESS attributed to GVHD.
13. Creatinine clearance < 30 mL/min calculated by Cockcroft-Gault equation.
14. Sodium (Na) concentration < 130 mmol/L.
15. Karnofsky Performance Status (KPS) or Lansky Performance Status < 20%.
16. Intensive care unit (ICU) care, life expectancy of less than 28 days, ongoing or unresolved hepatic sinusoidal obstruction syndrome, unstable hemodynamics, or evidence of current or previous clinically significant disease, medical condition or finding (including vital signs and ECG) that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.
17. History of allergy or hypersensitivity to any systemically administered antibody agent or its excipients.
18. Pregnancy or nursing.
19. Less than 12 years of age.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Neihulizumab - AUC | Up to Day 56
  Including AUC0-t, AUC0-tz, AUC 0-inf
Pharmacokinetics of Neihulizumab - Cmax | Up to Day 56
  Maximum plasma concentration
Pharmacokinetics of Neihulizumab - tmax | Up to Day 56
  Time to reach Cmax
Pharmacokinetics of Neihulizumab - Lambda-z | Up to Day 56
  Terminal phase elimination rate constant
Pharmacokinetics of Neihulizumab - t1/2 | Up to Day 56
  Half life
Pharmacokinetics of Neihulizumab - MRT | Up to Day 56
  Mean Residence Time
Pharmacokinetics of Neihulizumab - Vz and Vss | Up to Day 56
  Volume of distribution and volume of distribution at steady state

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to Day 180
  AEs graded according to CTCAE v4.03
To measure the Receptor Occupancy (RO) | Up to Day 56
  Receptor occupancy will be monitored using a flow cytometry based method
To measure regenerating islet-derived 3-alpha (REG3α) and suppression of tumorigenicity 2 (ST2) as Pharmacodynamics (PD) biomarkers. | Up to Day 56
  Receptor occupancy will be monitored using a flow cytometry based method
Complete Response (CR) | Day 28
  To assess the rate of complete response (CR) at Day 28 in patients treated with Neihulizumab
Overall Response Rate (ORR) | Day 28
  To assess the Overall Response Rate (ORR) at Day 28: CR+PR
Duration of Response | Up to Day 180
  For subjects with CR at Day 28, duration of response will be assessed according to the time interval from Day 28 to the first occurrence of (1) resumption of Neihulizumab administration or initiation of new systemic treatment for aGvHD or (for patients who have tapered steroids) an increase in corticosteroids to methylprednisolone 2 mg/kg (+/-10%) equivalent or more, or (2) death.
Non Relapse Mortality (NRM) | Day 180
  Patients will be followed-up for survival for 6 months after the first Neihulizumab treatment
Immunogenicity | Up to Day 56
  Immunogenicity will be monitored by anti-drug antibody (ADA) ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, PhD, Study Director — AltruBio, Inc. (formerly AbGenomics International); Paul Martin, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (13):
- United States (13):
  - City of Hope, Duarte, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Baylor College of Medicine-Houston Methodist & Texas Children's Hospital, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No